CLINICAL TRIAL: NCT01178424
Title: My Depression Wellness Toolkit Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Zindel Segal, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 093/2010
Record Dates: First submitted 2010-08-09; First posted 2010-08-10 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Major Depression
Keywords: Unipolar depression; Mindfulness based cognitive therapy; Cognitive behavioural Therapy; Functional magnetic resonance imaging; Relapse; Depressive relapse; Dysphoric; Cognitive reactivity; Serotonin transporter gene
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder; Recurrence | interventions — Mindfulness-Based Cognitive Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Based Cognitive Therapy (Experimental): Mindfulness Based Cognitive Therapy is a manualized, group skills training program (Segal et al., 2013) that is based on an integration of aspects of cognitive therapy for depression (Beck, 1979) with components of the mindfulness-based stress reduction program (Kabat-Zinn, 1990). Patients participate in 8 weekly sessions, each of which incorporates didactic and experiential learning, along with home practice of mindfulness skills taught in the program.
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy
- Cognitive Behaviour Therapy (Active Comparator): CBT is an evidence based depression-specific psychotherapy that examines the relationship between thinking styles and the perpetuation of mood symptoms in major depression. Patients use thought records and activity scheduling, among other tools, to record and reappraise their thinking during situations where negative affect is present, both in session and for homework.
  Interventions: Behavioral: Cognitive Behaviour Therapy

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy — Mindfulness-Based Cognitive Therapy, a manualized, group skills training program (Segal et al., 2013) that is based on an integration of aspects of cognitive therapy for depression (Beck, 1979) with components of the mindfulness-based stress reduction program (Kabat-Zinn, 1990). Patients participate in 8 weekly sessions, each of which incorporates didactic and experiential learning, along with home practice of skills taught in the program.
  Arms: Mindfulness Based Cognitive Therapy
Behavioral: Cognitive Behaviour Therapy — CBT is an evidence based depression-specific psychotherapy that examines the relationship between thinking styles and the perpetuation of mood symptoms in major depression. Patients use thought records and activity scheduling, among other tools, to record and reappraise their thinking during situations where negative affect is present, both in session and for homework.
  Arms: Cognitive Behaviour Therapy

SUMMARY:
Major depressive disorder (MDD) continues to have a profound impact on individuals, families, and the health care system. Despite marked success in treating active individual episodes of unipolar depression, our understanding of the neural and cognitive mechanisms involved in the return of symptoms remains extremely limited, and few interventions exist that specifically target factors involved in prophylaxis. The research being proposed is among the first that is designed to examine neurocognitive markers for depressive relapse vulnerability and link them directly to clinical prognosis.

Hypothesis 1: Cortical midline structures (CMS) network recruitment will be associated with behavioural and neural indices of a reflexive attentional bias towards dysphoric stimuli in a divided attention task.

Hypothesis 2: Behavioural and neural indices of dysphoric attentional bias following mood challenge will predict depression relapse in prospective 18-month follow up.

Hypothesis 3: Relative to CBT, Mindfulness Based Cognitive Therapy (MBCT) will normalize CMS and right insular/fronto-opercular cortices (INS-FO) network imbalance.

Hypothesis 4: Relative to CBT, MBCT will normalize to healthy control levels, behavioural and neural indices of dysphoric attentional bias, which will be predictive of reduced relapse risk across a 24 month follow up.

DETAILED DESCRIPTION:
Relapse and recurrence following recovery from Major Depressive Disorder (MDD) are common and debilitating outcomes that carry enormous social costs [1-3]. Our CIHR funded program of research has studied the nature of psychological vulnerability in affective disorder. We have recently identified the activation of a depressive cognitive mode triggered by temporary dysphoric states as a reliable risk marker for depressive relapse [4, see attached]. In parallel, functional imaging studies have increased our understanding of the neural mechanisms underlying normative affective responses [5] and have begun to examine their dysregulation in affective disorder [6-8]. Our research has identified potential brain biomarkers that predict episode relapse in unipolar depression. However, it remains unknown how these potential biomarkers are related to dysphoria-triggered information processing modes that also predict relapse, and whether these neurocognitive vulnerabilities are amenable to intervention, resulting in more lasting prophylaxis. The present proposal employs a cognitive neuroscience approach to examine whether our previously identified neural markers of depression relapse and prophylaxis are associated with a dysphoric information processing mode. In particular, we will use functional magnetic resonance imaging (fMRI) and behavioural probes to undertake a finely tuned examination of mood linked biases in attention toward dysphoric stimulus events (i.e., sad faces) to link our previously identified neural markers with a specific information processing mode. Further, our preliminary data presented here demonstrate a correlation between these mood linked neural markers and relapse, but we cannot demonstrate that these markers are causally related to relapse or prophylaxis. To address this, we will examine whether these markers and associated dysphoric attentional biases are 1) modifiable via attentional training designed to overcome reflexive modes of thought and perception and 2) are predictive of relapse status across an 24-month prospective follow up of treated patients. This research will elucidate the neural and information processing correlates that may signal relapse risk in recovered depressed patients. This knowledge will increase our limited understanding of the mechanisms underlying enduring depressive relapse vulnerability as well as assess potentially efficient strategies for relapse prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Women or men 18-65 years of age
* Meeting criteria for prior depression, currently in recovery or remission, according to Diagnostic and Statistical Manual of Mental Disorders (4th eg; DSM-IV-TR, (American Psychiatric Association, 2000)
* A baseline score of ≤ 12 on the HRSD (Hamilton, 1960)
* Internet access
* English proficiency at or above a grade 8 level

Exclusion Criteria:

* Schizophrenia or current psychosis
* Organic mental disorder
* Pervasive developmental delay (PDD)
* Current substance dependence
* Imminent suicide or homicide risk
* Axis I or II disorder that necessitates primary treatment not provided in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Rates of relapse/recurrence based on CMS and INS/FO configuration. | 2 years
  Patients who relapse will show Increased neural activation in CMS compared to INS/FO regions compared to non relapsers

SECONDARY OUTCOMES:
Changes in CMS and INSFO network imbalance following MBCT compared to CBT | 2 years
  Patients in MBCT will show greater levels of activation in INS/FO compared to patients in CBT
Changes in attentional processing of dysphoric stimuli between the groups | 8 weeks
  Relapsers will show greater attention to negative self-descriptive adjectives compared to non-relapsers.

CONTACTS AND LOCATIONS:
Overall Officials: Zindel V. Segal, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Background] Farb NA, Segal ZV, Mayberg H, Bean J, McKeon D, Fatima Z, Anderson AK. Attending to the present: mindfulness meditation reveals distinct neural modes of self-reference. Soc Cogn Affect Neurosci. 2007 Dec;2(4):313-22. doi: 10.1093/scan/nsm030. PMID 18985137
- [Background] Farb NA, Anderson AK, Mayberg H, Bean J, McKeon D, Segal ZV. Minding one's emotions: mindfulness training alters the neural expression of sadness. Emotion. 2010 Feb;10(1):25-33. doi: 10.1037/a0017151. PMID 20141299
- [Background] Segal ZV, Bieling P, Young T, MacQueen G, Cooke R, Martin L, Bloch R, Levitan RD. Antidepressant monotherapy vs sequential pharmacotherapy and mindfulness-based cognitive therapy, or placebo, for relapse prophylaxis in recurrent depression. Arch Gen Psychiatry. 2010 Dec;67(12):1256-64. doi: 10.1001/archgenpsychiatry.2010.168. PMID 21135325
- [Background] Segal, Z. V., Williams, J. M., & Teasdale, J. D. (2013). Mindfulness-based cognitive therapy for depression (2nd ed.). New York: Guilford Press.
- [Derived] Wu LC, Segal ZV, Farb NAS. Depression vulnerability and gray matter integrity of interoceptive networks in remitted depressed outpatients. J Affect Disord. 2025 Jul 1;380:113-123. doi: 10.1016/j.jad.2025.03.106. Epub 2025 Mar 21. PMID 40122253
- [Derived] Farb NAS, Desormeau P, Anderson AK, Segal ZV. Static and treatment-responsive brain biomarkers of depression relapse vulnerability following prophylactic psychotherapy: Evidence from a randomized control trial. Neuroimage Clin. 2022;34:102969. doi: 10.1016/j.nicl.2022.102969. Epub 2022 Feb 19. PMID 35367955
- [Derived] Segal ZV, Anderson AK, Gulamani T, Dinh Williams LA, Desormeau P, Ferguson A, Walsh K, Farb NAS. Practice of therapy acquired regulatory skills and depressive relapse/recurrence prophylaxis following cognitive therapy or mindfulness based cognitive therapy. J Consult Clin Psychol. 2019 Feb;87(2):161-170. doi: 10.1037/ccp0000351. Epub 2018 Nov 15. PMID 30431297
- [Derived] Farb N, Anderson A, Ravindran A, Hawley L, Irving J, Mancuso E, Gulamani T, Williams G, Ferguson A, Segal ZV. Prevention of relapse/recurrence in major depressive disorder with either mindfulness-based cognitive therapy or cognitive therapy. J Consult Clin Psychol. 2018 Feb;86(2):200-204. doi: 10.1037/ccp0000266. Epub 2017 Dec 21. PMID 29265831
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital. It is fully affiliated with the University of Toronto, and is a PAHO/WHO Collaborating Centre — http://www.camh.net/research